CLINICAL TRIAL: NCT03488277
Title: Evaluation of the Efficiency of Leg Elevation for Preventing Post Spinal Hypotension in Cesarean Section
Brief Title: Leg Elevation for Prevention of Post Spinal Hypotension in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of the anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Mater1
Record Dates: First submitted 2018-03-22; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Effects of; Anesthesia, Spinal and Epidural, in Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LE: leg elevation group (Experimental): the patients of this group will be positionned in supine with 15° left tilt and will have a leg elevation with a 30 cm pillow positionned under the heels. this position will be hold immediately after spinal anesthesia until fetal extraction
  Interventions: Other: leg elevation
- CG: Control group (No Intervention): The patients of this group will be positiooned in supine with 15° left tlit after spinal anesthesia. no leg elevation

INTERVENTIONS:
Other: leg elevation — intra operative position that consists in leg elevation with a 30 cm height pillow under the patient's heels
  Arms: LE: leg elevation group

SUMMARY:
Prospective trial including full term parturients scheduled for a cesarean section under spinal anesthesia. patients are being randomly assigned into 2 groups:

LE group: will be positioned in 15° left tilt with leg elevation with a 30cm height pillow under the heels, this position will be hold after spinal anesthesia until fetal extraction.

Control group: will be positioned in supine with 15° left tilt. the 2 groups will receive a 10ml/kg of crystalloid co-load intravenously, and the spinal anesthesia will be performed in sitting position with the same dose of Bupivacain, morphine and sufentanil.

DETAILED DESCRIPTION:
Prospective trial including full term parturients scheduled for a cesarean section under spinal anesthesia. patients are being randomly assigned into 2 groups:

LE group: will be positioned in 15° left tilt with leg elevation with a 30cm height pillow under the heels, this position will be hold after spinal anesthesia until fetal extraction.

Control group: will be positioned in supine with 15° left tilt. the 2 groups will receive a 10ml/kg of crystalloid co-load intravenously, and the spinal anesthesia will be performed in sitting position with the same dose of Bupivacain, morphine and sufentanil. we will record the demographic data, pre and intraoperative hemodynamic parameters, the dose of ephedrine required to treat post spinal hypotension and fetal parameters: pH and blood lactates

ELIGIBILITY:
Inclusion Criteria:

* full term parturients
* age> 18 Y
* scheduled of elective or urgent cesarean section under spinal anesthesia

Exclusion Criteria:

* patients who had general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post spinal hypotension | during the first 30minutes after the spinal anesthesia
  change of systolic blood pressure from baseline< 90 mmHg

SECONDARY OUTCOMES:
Lowest systolic blood pressure | during the first 30 minutes following spinal anesthesia
  the lowest systolic blood pressure observed after spinal anesthesia
ephedrine consumption | during the first 30 minutes following the spinal anesthesia
  total dose of Ephedrine received to treat post spinal hypotension
Fetal ph | 30 minutes after spinal anesthesia
  fetal ph measured with blood gas analysis
Fetal blood lactates | 30 minutes after spinal anesthesia
  fetal blood lactates (mmol/L) measured with blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami Mebazaa, Professor, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided